CLINICAL TRIAL: NCT01244633
Title: Ecopipam Treatment of Tourette Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Psyadon Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSY301
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-06

CONDITIONS: Tourette's Syndrome
Keywords: Tourette's; Ecopipam; Dopamine receptors; Efficacy; Safety; Adults
MeSH Terms: conditions — Tourette Syndrome | interventions — ecopipam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ecopipam (Experimental): Active treatment
  Interventions: Drug: Ecopipam

INTERVENTIONS:
Drug: Ecopipam — 50 or 100 mg tablets given once per day for eight weeks
  Other Names: SCH 39166; PSYRX 101

SUMMARY:
Tourette's Syndrome is a neurological disease characterized by verbal and motor tics. The currently available drug treatments are considered to be inadequate. This clinical trial is designed to test if ecopipam is effective for the treatment of Tourette's Syndrome in adults.

DETAILED DESCRIPTION:
Tourette's Syndrome is a neurological disease characterized by verbal and motor tics. Although its causes are unknown, many researchers believe that changes in brain chemicals (called neurotransmitters) are critically involved. One of these neurotransmitters is called dopamine, and it exerts its actions through its receptors (called D1-type or D2-type). It has been suggested that the symptoms of Tourette's Syndrome are due to an overactivity at the D1-type receptor. Ecopipam is a selective antagonist of the D1-type receptors. The present clinical trial is designed to test if ecopipam is able to relieve the symptoms of the disease in adults patients with Tourette's Syndrome. Eligible patients will be treated for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have TS (Tourette's Syndrome) based on the clinician-administered DCI (Diagnostic Confidence Index) for TS.
* Subjects must exhibit both motor and vocal tics.
* Subjects must have exhibited tics for >5 years.
* Subjects must have a minimum score of 20 at both Screening and Baseline (just prior to the first treatment) on the YGTSS (Yale Global Tic Severity Score).
* Subjects must be age ≥ 18 years.
* Women must be postmenopausal (> 12 months without menses) or surgically sterile (i.e., by hysterectomy and/or bilateral oophorectomy) or must be using effective contraception (i.e., oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for the duration of their participation in the study. Women of childbearing potential must agree to use contraception for 30 days after their last dose of study drug.
* Sexually active male subjects must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of study drug.
* Subject must execute a written informed consent.

Exclusion Criteria:

* Subjects who have unstable medical illness or clinically significant abnormalities on laboratory tests, or ECG at Screening.
* Subjects with a major depressive episode in the past 2 years
* Subjects with a history of attempted suicide
* Subjects with clinically significant suicidality (score of ≥ 2 on Item 3 for the Hamilton Depression Rating Scale [HAM-D])
* Subjects with a first-degree relative with a major depressive episode that resulted in any psychiatric hospitalization, attempted or completed suicide
* Subjects with a history of seizures.
* Subjects with a myocardial infarction within 6 months.
* Women of childbearing potential who are currently pregnant or lactating.
* Subjects who have a need for medication (other than ecopipam) with possible effects on TS symptoms (i.e., lithium, naltrexone, methylphenidate, or psychostimulants), unfavorable interactions with ecopipam (ie, dopamine agonists [including bupropion]), or monoamine oxidase inhibitors.
* Subjects with a lifetime history of bipolar disorder type I or II, dementia, schizophrenia, or any psychotic disorder determined by the Structured Clinical Interview for Diagnostic Statistical Manual IV Text Revision (DSM-IV-TR) Axis-I Disorders (SCID).
* Subjects with current or recent (past 3 months) DSM-IV substance abuse or dependence (with the exception of nicotine).
* Subjects with positive urine drug screen (cocaine, amphetamine, methamphetamine, tetrahydrocannabinol (THC), benzodiazepines, barbiturates, phencyclidine (PCP), opiates) at Screening. Subjects with urine positive only for benzodiazepines and/or marijuana (i.e., a user but not an abuser as based on DSM-IV criteria) may be eligible.
* Subjects who have had previous treatment with ecopipam.
* Subjects who have had treatment with:

  * investigational medication or depot neuroleptics within 3 months
  * fluoxetine within 6 weeks
  * other psychotropics with possible effects on TS symptoms (ie, lithium, or naltrexone) within 2 weeks prior to Screening.
  * oral neuroleptics within 2 weeks
  * selective serotonin reuptake inhibitors unless the dosage has been stable for a minimum of 4 weeks prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Gilbert, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Atlantic Neuroscience Institute Overlook Hospital, Summit, New Jersey
  - North Shore Hospital, Manhasset, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Background] Chipkin RE, Iorio LC, Coffin VL, McQuade RD, Berger JG, Barnett A. Pharmacological profile of SCH39166: a dopamine D1 selective benzonaphthazepine with potential antipsychotic activity. J Pharmacol Exp Ther. 1988 Dec;247(3):1093-102. PMID 2905002
- See also: Link to Sponsor's Website — http://www.psyadonrx.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ecopipam
Started | 18
Completed | 15
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ecopipam
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Yale Global Tic Severity Score
Description: The Yale Global Tic Severity Score is a composite of subject reported severity of motor (range 0-25) and vocal (range 0-25) tics , as well as an impairment score (range 0-50). The outcome we are using is the Total Tic Severity score which is the sum of the motor and vocal tic severity scores (range 0-50). The higher the score on this scale, the more severe the symptoms. A positive drug effect is associated with a decrease from baseline.
Time Frame: 8 weeks
Population: Subjects completing the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ecopipam
Number analyzed (Participants) | 15
units on a scale | 25.3 (9.2)

2. Secondary Outcome: Adult Attention Deficit/Hyperactivity Disorder (ADHD) Self-report Symptom Checklist (ASRS)
Description: This is a standard measure of ADHD severity that is typically used in these types of clinical trials.
Time Frame: Every 7 days
Reporting Status: Not Posted

3. Secondary Outcome: Hamilton Depression Scale
Description: This is a measure of feelings of depression that the patient might have.
Time Frame: Every 7 days
Reporting Status: Not Posted

4. Secondary Outcome: Premonitory Urge for Tics Scale (PUTS-1)
Description: This is a measure of the tic behavior that is seen in Tourette's patients, and it is typically used in these types of trials.
Time Frame: Every 7 days
Reporting Status: Not Posted

5. Secondary Outcome: Clinician Global Impression - Improvement and Severity Scales (CGI)
Description: This is a measure of how the treating physician perceives the effectiveness of a drug treatment, and it is typically used in these types of clinical trials.
Time Frame: End of trial
Reporting Status: Not Posted

6. Secondary Outcome: Safety Assessments
Description: Patients will be evaluated for any adverse events, and they will have a variety of blood tests to examine if any changes occur.
Time Frame: Every 7 days
Reporting Status: Not Posted

7. Secondary Outcome: Columbia Scale for Suicide Risk
Description: This test monitors whether the patient has any feelings of committing self-harm. It is mandated by the FDA to include this scale in all clinical trials of new central nervous system drugs.
Time Frame: Every 7 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Ecopipam
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ecopipam (N=18)
Insomnia (Nervous system disorders) | 6

LIMITATIONS AND CAVEATS:
This was an open label study with no placebo control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No